CLINICAL TRIAL: NCT03642340
Title: A Post-marketing Surveillance to Assess Safety and Efficacy of Besivo
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: ID-BSB-401
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a post-marketing surveillance of Besivo in participants with chronic hepatitis B.

DETAILED DESCRIPTION:
This post-marketing surveillance required by Korea MFDS regulation. The objectives of this study are to monitor adverse events and effectiveness of Besivo.

ELIGIBILITY:
Inclusion Criteria:

* The patient diagnosed with chronic hepatitis B.
* The patient who is first prescribed and administered Besivo.

Exclusion Criteria:

* The patients who are overreacting to this drug or its components
* Medium to severe Renal function disorder
* The patient under 19
* The Patient who are taboo with L-Carnitine

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 3000
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-05-15 (Actual); Primary Completion 2023-05-14 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse event after this drug administration in general medical practice. | 48weeks
  Any adverse events occurred after this drug dosing will be recorded. Description of adverse event(s) including type of adverse event(s), onset/end date, severity, action taken, causal relationship to the drug and investigator's view on the adverse event(s) will be captured, whether it is related to the drug or not and until follow up visit more than 1 time during the surveillance period.
  Lab abnormalities and changes in vital signs are considered to be adverse events only if they result in discontinuation from the study, necessitate therapeutic medical intervention, and/or if the investigator considers them to be adverse events.
Incidence of serious adverse event after this drug administration in general medical practice. | 48 weeks
  Any serious adverse events occurred after this drug dosing will be recorded. Description of serious adverse event(s) including type of serious adverse event(s), onset/end date, severity, action taken, causal relationship to the drug and investigator's view on the serious adverse event(s) will be captured, whether it is related to the drug or not and until follow up visit more than 1 time during the surveillance period.
  Lab abnormalities and changes in vital signs are considered to be adverse events only if they result in discontinuation from the study, necessitate therapeutic medical intervention, and/or if the investigator considers them to be adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Ildong Ildong, Study Director — PV
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided